CLINICAL TRIAL: NCT00985114
Title: An Open Label, Randomized, Controlled Study of a Second Generation EndoBarrier™ Liner vs. Diet Control for the Treatment of Type 2 Diabetes
Brief Title: Safety and Efficacy Study of EndoBarrier in Subjects With Type II Diabetes and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-1
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Type II Diabetes
Keywords: Type II Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device (Experimental): EndoBarrier implanted for 6 months. Subject followed for 6 months after device was explanted.
  Interventions: Device: EndoBarrier; Behavioral: Diet + Lifestyle Counseling
- Diet + Lifestyle counseling (Active Comparator): Multidisciplinary lifestyle and nutritional counseling for 12 months
  Interventions: Behavioral: Diet + Lifestyle Counseling

INTERVENTIONS:
Device: EndoBarrier — EndoBarrier implant
  Arms: Device
Behavioral: Diet + Lifestyle Counseling — Multidisciplinary lifestyle and nutritional counseling

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a second generation EndoBarrier Liner compared to a study diet to treat Subjects with Type 2 Diabetes.

This is a randomized, controlled study which will enroll approximately 70 Subjects with Type 2 Diabetes. Randomization will be one to one with approximately 35 EndoBarrier device Subjects and approximately 35 study diet Subjects. Subjects randomized as diet Subjects will be offered the EndoBarrier device after 12 months on study at the investigator's discretion if treatment of the device subjects indicates adequate efficacy. This study will be conducted at three (3) investigational sites.

The primary efficacy endpoint is:

* Assessment of the percent (%) of Subjects who achieve a ≥ 0.5% reduction in HbA1C at 24 weeks or last visit from baseline between the two groups.

Secondary endpoints are:

* Percent (%) of Subjects who achieve a HbA1C of 7.0% or lower at week 24 or last visit from baseline.
* Percent (%) of Subjects who have their diabetic medication(s) dosage decreased or discontinued at week 24 or last visit from baseline.
* Percent (%) of Subjects who achieve a decrease in post-prandial excursions as evidenced by challenge to a standardized meal tolerance test (MTT) at week 24 or last visit from baseline.
* Assessment of absolute weight loss (Kg) at week 24 or last visit from baseline.
* Percent (%) of Subjects who maintain a HbA1c lower than their baseline assessment at 12 months.
* Compare physical component summary (PCS), mental component summary (MCS) and quality adjusted life years (QALYs)via analysis of the SF-36v2 QOL.

DETAILED DESCRIPTION:
Utilization of the EndoBarrier Gastrointestinal Liner in obese subjects with T2DM demonstrated an acceptable safety profile with clinically significant improvements in glycemic control and body weight when compared to a similar diet controlled group of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 65 years
* Male or Female
* Subjects with Type 2 Diabetes who have been treated for ≤10 years
* BMI> 30 - < 50
* Subjects with an HbA1c level > 7.5 and ≤ 10.0%
* Subjects taking a combination of metformin and sulfonylureas and/or insulin (other than pre-mixed long and short acting insulins, ie. NovoMix 30)
* Patients willing to comply with study requirements
* Patients who have signed an informed consent form

Exclusion Criteria:

* Subjects taking oral medications to control their diabetes other than sulfonylureas and metformin
* Subjects diagnosed with Type 1 Diabetes Mellitus or having a history of ketoacidosis
* Subjects on insulin > 10 years
* Subjects requiring insulin > 70 units per day
* Subjects on pre-mixed insulin (ie. NovoMix 30)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Greve, MD, Principal Investigator — University Hospital Masstricht
Locations (3):
- Netherlands (3):
  - Ziekenhuis Rijnstate Arnhem, Arnhem
  - Medisch Centrum Parkstad, Heerlen
  - University Hospital Maastricht, Maastricht

IPD SHARING:
Plan to Share IPD: Undecided
Yes
  De-identified individual subject data is on file at the Sponsor

REFERENCES:
- [Derived] de Jonge C, Rensen SS, Verdam FJ, Vincent RP, Bloom SR, Buurman WA, le Roux CW, Bouvy ND, Greve JW. Impact of Duodenal-Jejunal Exclusion on Satiety Hormones. Obes Surg. 2016 Mar;26(3):672-8. doi: 10.1007/s11695-015-1889-y. PMID 26446491
- [Derived] Koehestanie P, de Jonge C, Berends FJ, Janssen IM, Bouvy ND, Greve JW. The effect of the endoscopic duodenal-jejunal bypass liner on obesity and type 2 diabetes mellitus, a multicenter randomized controlled trial. Ann Surg. 2014 Dec;260(6):984-92. doi: 10.1097/SLA.0000000000000794. PMID 25072436
- [Derived] de Jonge C, Rensen SS, Koek GH, Joosten MF, Buurman WA, Bouvy ND, Greve JW. Endoscopic duodenal-jejunal bypass liner rapidly improves plasma parameters of nonalcoholic fatty liver disease. Clin Gastroenterol Hepatol. 2013 Nov;11(11):1517-20. doi: 10.1016/j.cgh.2013.07.029. Epub 2013 Aug 3. PMID 23920034

RESULTS

PARTICIPANT FLOW:
Groups:
- EndoBarrier Device: EndoBarrier
  EndoBarrier: EndoBarrier implant
Period: Overall Study
Arm/Group | EndoBarrier Device | Diet + Lifestyle Counseling
Started | 34 (38 randomized, 34 received the device) | 39
Diet + Lifestyle Counseling Cross-over | 0 | 28 (Received device for intended period of 12 months with 6 months follow up)
Completed | 33 | 37
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Device: EndoBarrier
  EndoBarrier: EndoBarrier implant
- Total: Total of all reporting groups
Arm/Group | Device | Diet + Lifestyle Counseling | Total
Number analyzed (Participants) | 34 | 39 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (9.1) | 49.3 (7.8) | 49.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 21 | 25 | 46
Region of Enrollment [Number; unit: participants]
  Netherlands | 34 | 39 | 73
Baseline weight [Mean (Standard Deviation); unit: kg] | 110.1 (19.5) | 113.5 (19.3) | 111.9 (19.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent (%) of Subjects Who Achieve a ≥ 0.5% Reduction in HbA1C at 24 Weeks or Last Visit From Baseline.
Time Frame: 6 months
Measure: Number; unit: % of participants
Arm/Group | Device | Diet + Lifestyle Counseling
Number analyzed (Participants) | 33 | 36
% of participants | 81.8 | 61.1

ADVERSE EVENTS:
Groups:
- Device and Cross Over: EndoBarrier
  EndoBarrier: EndoBarrier implant
Arm/Group | Device and Cross Over | Diet + Lifestyle Counseling
Serious Adverse Events (participants affected / at risk) | 18/66 | 4/39
Other Adverse Events (participants affected / at risk) | 55/66 | 25/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device and Cross Over (N=66) | Diet + Lifestyle Counseling (N=39)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Kidney carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Scapula fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute hernia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pylorospasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Procedural Nausea (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural Vomiting (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device and Cross Over (N=66) | Diet + Lifestyle Counseling (N=39)
Abdominal pain upper (Gastrointestinal disorders) | 31 (47) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 11 (15) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 13 (20) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (15) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 14 (21) | 6 (6)
Vomiting (Gastrointestinal disorders) | 8 (11) | 4 (4)
Procedural nausea (Injury, poisoning and procedural complications) | 17 (18) | 0 (0)
Procedural vomiting (Gastrointestinal disorders) | 8 (8) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 14 (48) | 11 (11)
Hypovitaminosis (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 18 (22) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia (Infections and infestations) | 1 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No